CLINICAL TRIAL: NCT03939624
Title: Sodium-glucose Cotransporter 2 (SGLT2) Inhibitors and the Risk of Cardiovascular Events Among Patients with Type 2 Diabetes: a Multicenter Cohort Study
Brief Title: Sodium-glucose Cotransporter 2 (SGLT2) Inhibitors and Risk of Cardiovascular Events
Status: Completed | Type: Observational
Sponsor: Canadian Network for Observational Drug Effect Studies, CNODES (Other)
Collaborators: Drug Safety and Effectiveness Network, Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: Q18-06
Record Dates: First submitted 2019-05-03; First posted 2019-05-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-01

CONDITIONS: Type2 Diabetes; Myocardial Infarction; Ischemic Stroke; Cardiovascular Death; Heart Failure; All-Cause Mortality
Keywords: Sodium-Glucose Cotransporter 2 Inhibitors; Type 2 Diabetes; Myocardial Infarction; Ischemic Stroke; Cardiovascular Death
MeSH Terms: conditions — Myocardial Infarction; Ischemic Stroke; Heart Failure; Diabetes Mellitus, Type 2 | interventions — Sodium-Glucose Transporter 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Sodium-glucose cotransporter 2 (SGLT2) inhibitors: Patients who received a SGLT2 inhibitor alone (canagliflozin, dapagliflozin, empagliflozin) or in combination with non-DPP4 inhibitor drugs at cohort entry date.
  Interventions: Drug: Sodium-glucose cotransporter 2 (SGLT2) inhibitors
- Dipeptidyl peptidase-4 (DPP-4) inhibitors: Patients who received a DPP-4 inhibitor (alogliptin, linagliptin, saxagliptin, sitagliptin, vildagliptin) alone or in combination with non-SGLT2 inhibitor drugs at cohort entry date.
  Interventions: Drug: Dipeptidyl peptidase-4 (DPP-4) inhibitors

INTERVENTIONS:
Drug: Sodium-glucose cotransporter 2 (SGLT2) inhibitors — Exposure to SGLT2 will be defined as a prescription for a SGLT2 inhibitor alone (canagliflozin, dapagliflozin, empagliflozin) or in combination with non-DPP4 inhibitor drugs at cohort entry date.
  Other Names: ATC A10BK, A10BD15, A10BD16, A10BD19, A10BD20, A10BD21, A10BD23, A10BD24, A10BD25
  Groups: Sodium-glucose cotransporter 2 (SGLT2) inhibitors
Drug: Dipeptidyl peptidase-4 (DPP-4) inhibitors — Exposure to DPP-4 will be defined as a prescription for a DPP-4 inhibitor (alogliptin, linagliptin, saxagliptin, sitagliptin, vildagliptin) alone or in combination with non-SGLT2 inhibitor drugs at cohort entry date.
  Other Names: ATC A10BH, A10BD07, A10BD08, A10BD09, A10BD10, A10BD11, A10BD12, A10BD13, A10BD18, A10BD19, A10BD20, A10BD21, A10BD22, A10BD24, A10BD25
  Groups: Dipeptidyl peptidase-4 (DPP-4) inhibitors

SUMMARY:
The purpose of this study is to compare the risk of cardiovascular events associated with the use of sodium-glucose cotransporter 2 (SGLT2) inhibitors in comparison with the use of dipeptidyl peptidase-4 (DPP-4) inhibitors among patients with type 2 diabetes.

The investigators will carry out separate population-based cohort studies using health care databases in seven Canadian provinces and the United Kingdom. The study cohort will be defined by the initiation of a SGLT2 inhibitor or a DPP-4 inhibitor after SGLT2 inhibitors entered the market. Patients will be followed up until the occurrence of a cardiovascular event. The results from the separate sites will be combined by meta-analysis to provide an overall assessment of the risk of cardiovascular events in users of SGLT2 inhibitors.

The investigators hypothesize that the use of SGLT2 inhibitors will be associated with a decreased risk of cardiovascular events in comparison with the use of DPP-4 inhibitors.

DETAILED DESCRIPTION:
The objective of this study is to compare the risk of major adverse cardiac events (MACE) associated with the use of sodium-glucose cotransporter 2 (SGLT2) inhibitors in comparison with the use of dipeptidyl peptidase-4 (DPP-4) inhibitors among patients with type 2 diabetes.

A common-protocol approach will be used to conduct retrospective cohort studies using administrative health care data from seven Canadian provinces (Alberta, British Columbia, Manitoba, Nova Scotia, Ontario, Quebec, and Saskatchewan) and the United Kingdom (UK) Clinical Practice Research Datalink (CPRD). Briefly, the Canadian databases include population-level data on physician billing, diagnoses and procedures from hospital discharge abstracts, and dispensations for prescription drugs. The data in Ontario will be restricted to patients aged 65 years old and older. The CPRD is a clinical database that is representative of the UK population and contains the records for patients seen at over 680 general practitioner practices in the UK; these data will be linked to the Hospital Episode Statistics (HES) database, which contains in-hospital diagnosis and procedure data.

The investigators will use a prevalent new-user cohort design (Suissa et al., 2017). In each jurisdiction, the investigators will assemble a source population that includes all patients who received an antidiabetic medication (metformin, sulfonylureas, thiazolidinediones, DPP-4 inhibitors, SGLT2 inhibitors, GLP-1 receptor agonists, alpha-glucosidase inhibitors, meglitinides, insulin, or combinations of these drugs) between January 1, 2006 and June 30, 2018 (or the latest date of data availability at each site). From this source population, a study cohort including all patients who received a prescription for a SGLT2 inhibitor or DPP-4 inhibitor on or after the date of the first dispensing (or prescription in CPRD) of a SGLT2 inhibitor in each jurisdiction and on or before June 30, 2018 (or latest date of data availability at each site) will be created. Study cohort entry date will be defined by the SGLT2 dispensation date or the corresponding dispensation date for a DPP-4 inhibitor in the matched exposure set. Patients will be followed until the occurrence of an event (defined below), death, end of healthcare coverage (plus 30 days), or end of the study period, whichever occurs first. Patients will be eligible to enter the cohort twice, a first time with a DPP-4 prescription and a second time with a SGLT2 prescription.

Exposure will be defined as a prescription for a SGLT2 inhibitor or a DPP-4 inhibitor on the date of cohort entry. DPP-4 inhibitors will serve as the reference category as both classes are second- to third-line therapy, and DPP-4 inhibitors have no known association with the outcome. Analyses will be conducted using an as-treated approach. Patients will be followed until drug discontinuation or the initiation of the other study drug. The primary outcome will be MACE, defined as a composite endpoint of myocardial infarction, ischemic stroke, or cardiovascular death. Secondary outcomes will include the individual endpoints of MACE, all-cause mortality, and hospitalization for heart failure.

Using a prevalent new-user design with time-based exposure sets, each user of a SGLT2 inhibitor will be matched to a DPP-4 inhibitor user on the number of prior antidiabetic medication classes and on time-conditional propensity score. Cox proportional hazards models will be used to estimate site-specific adjusted hazards ratios (HR) and corresponding 95% confidential intervals (CI) for each outcome of interest among patients exposed to a SGLT2 inhibitor in comparison to those exposed to a DPP-4 inhibitor. As secondary analyses, the MACE and heart failure outcomes will be stratified by age (≥70 and <70 years), sex, prior insulin use, and SGLT2 molecule. The MACE composite outcome will be stratified by history of cardiovascular disease, and the heart failure outcome by history of heart failure. Sensitivity analyses will be performed to assess the robustness of study results and address some of the study limitations. Meta-analyses of the site-specific results will be performed using random effects models.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received a prescription for a SGLT2 inhibitor or DPP-4 inhibitor on or after the date of the first dispensation of a SGLT2 inhibitor at each site and on or before June 30, 2018 (or latest date of data availability at each site)

Exclusion Criteria:

* Patients who received both a first prescription for a SGLT2 inhibitor and a DPP-4 inhibitor on the same date
* Patients with missing sex
* Patients aged less than 18 years at cohort entry date (<19 years in Alberta and <66 years in Ontario)
* Patients with less than 365 days of healthcare coverage prior to cohort entry date
* Patients with date inconsistencies or no follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In each jurisdiction, the investigators will assemble a source population that includes all patients who received an antidiabetic medication between January 1, 2006 and June 30, 2018. From this source population, a study cohort will be formed including all patients who received a prescription for a SGLT2 inhibitor or DPP-4 inhibitor on or after the date of the first dispensation of a SGLT2 inhibitor in each jurisdiction and on or before June 30, 2018. Study cohort entry date will be defined by the SGLT2 dispensation date or the corresponding dispensation date for a DPP-4 inhibitor in the matched exposure set.
Sampling Method: Probability Sample
Enrollment: 419734 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Myocardial infarction | Patients will be followed from the date of study cohort entry until hospitalization for myocardial infarction, treatment discontinuation, death, end of healthcare coverage, or for up to 64 months, whichever occurs first.
  Patients hospitalized for myocardial infarction recorded as the most responsible diagnosis or present on admission in the hospitalization record with the following ICD-10-CA codes: I21.x.
Ischemic stroke | Patients will be followed from the date of study cohort entry until hospitalization for ischemic stroke, treatment discontinuation, death, end of healthcare coverage, or for up to 64 months, whichever occurs first.
  Patients hospitalized for ischemic stroke recorded as the most responsible diagnosis or present on admission in the hospitalization record with the following ICD-10-CA codes: I63.x, I64.x.
Cardiovascular death | Patients will be followed from the date of study cohort entry until death, treatment discontinuation, end of healthcare coverage, or for up to 64 months, whichever occurs first.
  Cardiovascular death will be defined using the following algorithm:
  * In-hospital death with a cardiovascular diagnosis (ICD-10-CA: I00.x-I77.x (except I46.9)) recorded as the most responsible diagnosis or present on admission; or
  * Out-of-hospital death (including death in the emergency department) without:
    * Documentation of cancer (ICD-9-CM: 140-172, 174-209; ICD-10-CA: C00-C43, C45-C97) in hospital, emergency department or physician claims data in the prior year; or
    * Documentation of trauma (ICD-9-CM: 800-999, E000-E999; ICD-10-CA: S00-T98, V01-Y98) in hospital, emergency department or physician claims data in the preceding month.
  In a sensitivity analysis, the algorithm will be validated in the sites with access to vital statistics data with cause of death.

SECONDARY OUTCOMES:
All-cause mortality | Patients will be followed from the date of study cohort entry until death, treatment discontinuation, end of healthcare coverage, or for up to 64 months, whichever occurs first.
Heart failure | Patients will be followed from the date of study cohort entry until hospitalization for heart failure, treatment discontinuation, death, end of healthcare coverage, or for up to 64 months, whichever occurs first.
  Patients hospitalized for heart failure recorded as the most responsible diagnosis in the hospitalization record with the following ICD-10-CA codes: I11.0, I13.0, I13.2, I50.x.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Ernst, MD, MSc, FRCPC, Principal Investigator — Lady Davis Institute for Medical Research, Jewish General Hospital
Locations (1):
- Lady Davis Institute for Medical Research, Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brunetti VC, St-Jean A, Dell'Aniello S, Fisher A, Yu OHY, Bugden SC, Daigle JM, Hu N, Alessi-Severini S, Shah BR, Ronksley PE, Lix LM, Ernst P, Filion KB; Canadian Network for Observational Drug Effect Studies (CNODES) Investigators. Characteristics of new users of recent antidiabetic drugs in Canada and the United Kingdom. BMC Endocr Disord. 2022 Sep 29;22(1):241. doi: 10.1186/s12902-022-01140-1. PMID 36175881
- [Background] Suissa S, Moodie EE, Dell'Aniello S. Prevalent new-user cohort designs for comparative drug effect studies by time-conditional propensity scores. Pharmacoepidemiol Drug Saf. 2017 Apr;26(4):459-468. doi: 10.1002/pds.4107. Epub 2016 Sep 9. PMID 27610604
- [Background] Filion KB, Lix LM, Yu OH, Dell'Aniello S, Douros A, Shah BR, St-Jean A, Fisher A, Tremblay E, Bugden SC, Alessi-Severini S, Ronksley PE, Hu N, Dormuth CR, Ernst P, Suissa S; Canadian Network for Observational Drug Effect Studies (CNODES) Investigators. Sodium glucose cotransporter 2 inhibitors and risk of major adverse cardiovascular events: multi-database retrospective cohort study. BMJ. 2020 Sep 23;370:m3342. doi: 10.1136/bmj.m3342. PMID 32967856
- [Background] Lix LM, Sobhan S, St-Jean A, Daigle JM, Fisher A, Yu OHY, Dell'Aniello S, Hu N, Bugden SC, Shah BR, Ronksley PE, Alessi-Severini S, Douros A, Ernst P, Filion KB. Validity of an algorithm to identify cardiovascular deaths from administrative health records: a multi-database population-based cohort study. BMC Health Serv Res. 2021 Jul 31;21(1):758. doi: 10.1186/s12913-021-06762-0. PMID 34332563
- See also: This is the website describing the general functions of the organization, other CNODES projects, and investigator profiles. — http://www.cnodes.ca